CLINICAL TRIAL: NCT01366183
Title: Chemotherapy Toxicity in Elderly Women With Ovarian, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Chemotherapy Toxicity On Quality of Life in Older Patients With Stage I, Stage II, Stage III, or Stage IV Ovarian Epithelial, Primary Peritoneal Cavity, or Fallopian Tube Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0273; NCI-2011-02900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0273 (Other: Gynecologic Oncology Group); GOG-0273 (Other: DCP); GOG-0273 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Stage I Ovarian Cancer AJCC v6 and v7; Stage IA Fallopian Tube Cancer AJCC v6 and v7; Stage IB Fallopian Tube Cancer AJCC v6 and v7; Stage IC Fallopian Tube Cancer AJCC v6 and v7; Stage II Ovarian Cancer AJCC v6 and v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin; Filgrastim; Granulocyte Colony-Stimulating Factor; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (quality of life questionnaire): Patients receive chemotherapy comprising carboplatin, paclitaxel, and filgrastim (regimen 1) or carboplatin alone (regimen 2) every 21 days for 4 courses according to their physicians and/or patients' choice. Patients may undergo surgery and/or further chemotherapy at the discretion of treating physician. Patients undergo blood sample collection at baseline and periodically during course 1 for pharmacokinetic studies.
  Patients' quality of life is assessed by the FACT-O, the FACT-Ntx subscale, the IADL, and the Ability to Complete Social Activity questionnaires at baseline, prior to courses 1 and 3, and then 3-6 weeks after completion of course 4. Nutritional status, such as body mass index and weight loss, and comorbidity and hearing impairment are also assessed.
  Interventions: Procedure: Assessment of Therapy Complications; Drug: Carboplatin; Biological: Filgrastim; Drug: Paclitaxel; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Assessment of Therapy Complications — Undergo nutritional status, such as body mass index and weight loss, and comorbidity and hearing impairment assessments
Drug: Carboplatin — Undergo chemotherapy
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Filgrastim — Undergo chemotherapy
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Paclitaxel — Undergo chemotherapy
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the chemotherapy toxicity on quality of life in older patients with stage I, stage II, stage III, or stage IV ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer. Learning about the side effects of chemotherapy in older patients may help doctors plan better ways to treat cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To determine whether the score on Instrumental Activities of Daily Living (IADL) obtained prior to treatment is associated with the ability of patients to complete four cycles of chemotherapy without dose reduction or a more than 7-day delay.

II. To estimate by regimen the percentage of patients who are able to complete four cycles of chemotherapy regardless of dose reductions and delays.

III. To compare actual and calculated carboplatin area under the curve (AUC) in this patient population.

SECONDARY OBJECTIVES:

I. To describe the percentage of patients who are entered after primary surgery versus those entered to receive primary or neoadjuvant chemotherapy, the percentage of patients who are treated with each allowed regimen, and the percentage of patients who eventually receive surgery in the primary chemotherapy group.

II. To determine whether the need for assistance with IADLs at time of registration is associated with choice of chemotherapy regimen (in both primary chemotherapy and primary surgery patients).

III. To explore whether age, baseline scores on the geriatric measures (functional status, nutritional status, or co-morbidity) and quality-of-life (QOL) are correlated with likelihood of completing four courses of chemotherapy without dose reduction or a more than 7-day delay.

IV. To explore reasons for and timing of dose reductions and delays. V. To describe toxicities, pre-/post-chemotherapy QOL, and pre-/post-chemotherapy scores on geriatric measures in this patient population.

TERTIARY OBJECTIVES:

I. To explore potential relationships of carboplatin AUC, paclitaxel clearance, and paclitaxel time above a plasma concentration of 0.05 mcM to nadir neutrophil and platelet counts during course 1 of treatment.

II. To explore the association between baseline IADL and survival. III. To explore the association between IADL and the functional well-being (FWB) subscale in the Functional Assessment of Cancer Therapy ? Ovary (FACT-O).

OUTLINE:

Patients receive chemotherapy comprising carboplatin, paclitaxel, and filgrastim (regimen 1) or carboplatin alone (regimen 2) every 21 days for 4 courses according to their physicians and/or patients' choice. Patients may undergo surgery and/or further chemotherapy at the discretion of treating physician. Patients undergo blood sample collection at baseline and periodically during course 1 for pharmacokinetic studies.

Patients' quality of life is assessed by the FACT-O, the Functional Assessment of Cancer Treatment ? Neurotoxicity (FACT-Ntx subscale), the IADL, and the Ability to Complete Social Activity questionnaires at baseline, prior to courses 1 and 3, and then 3-6 weeks after completion of course 4. Nutritional status, such as body mass index and weight loss, and comorbidity and hearing impairment are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must have a histologically or cytologically confirmed diagnosis of adenocarcinoma of the ovary, peritoneum, or fallopian tube either by surgery, biopsy, fine-needle aspiration (FNA), paracentesis, or thoracentesis; a diagnosis of a mucinous cancer must be made by biopsy only
* International Federation of Gynecology and Obstetrics (FIGO) stage I, II, III, and IV are eligible
* Patients must have received no previous treatment for this malignancy other than surgery
* Patients must be entered within eight weeks of confirmation of disease diagnosis by surgery, biopsy, FNA, paracentesis or thoracentesis if there is no primary surgery, and within twelve weeks of primary or staging surgery if patient received primary surgery
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Bilirubin less than or equal upper limit of normal (ULN)
* Creatinine less than or equal to 1.5 x ULN
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, 2 or 3
* Effective XX/XX/2014, only patients 75 years of age or older are eligible for enrollment; (04/23/2012) (08/12/2013)
* Patients must have recovered from the effects of recent surgery
* Patients must be free of active infection requiring antibiotics
* Patients must have signed an approved informed consent and Health Insurance Portability and Accountability Act (HIPAA)
* Patient and physician agree that they plan to conduct treatment according to Regimen 3
* Patient can read and understand sufficient English to be able to respond to questions posed by the study instruments

Exclusion Criteria:

* Patients who have received previous treatment for this malignancy other than surgery
* Patients with other invasive malignancies whose previous cancer treatment contraindicates this protocol therapy
* ?Borderline tumors? (tumors of low malignant potential) by surgery or biopsy are excluded
* Patients with medical conditions that in the opinion of the investigator render treatment on this protocol unsafe should be excluded

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2011-08-15 (Actual); Primary Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerance to study treatment, defined as completing four cycles of study treatment, without dose reductions or treatment delays of over seven days | Up to 5 years
  Will be modeled with logistic regression using baseline IADL scores as a covariate. Exploratory analysis will evaluate baseline IADL scores adjusting for covariates such as: Charlson scale, nutritional status, or age.
Percent of women, who are 70 years or older, able to complete at least 4 cycles of treatment regardless of dose reduction and delays | Up to 5 years
  While this percentage will be estimated for each study regimen separately, the targeted sample size will limit the width of the 95%-confidence interval for the marginal percentage so that it is no larger than 0.15.

SECONDARY OUTCOMES:
Changes in quality-of-life measured by FACT-O, FACT/GOG-Ntx-4 subscale, IADL, and ADL | Baseline to up to 6 weeks after completion of course 4
  The changes in FACT-O, FACT/GOG-Ntx-4 subscale, IADL, and ADL will be summarized descriptively as the differences of scores between pre and post chemotherapy. Assuming 80% of patients complete the assessment at the completion of chemotherapy, then a sample of 148 patients will provide 90% power to detect 5 unit changes in FACT-O, 0.5 unit change in FACT/GOG-Ntx subscale score, 1 unit change in IADL or ADL score using paired t-test at significant level of 0.05.
Changes in comorbidity index measured by the Charlson scale | Baseline to up to 6 weeks after completion of course 4
Changes in nutritional status measured by weight | Baseline to up to 6 weeks after completion of course 4
  The changes in weight will be summarized descriptively as the differences of scores between pre and post chemotherapy. The change of nutritional status after completing chemotherapy will be examined using McNemar?s test.
Clinical response of elderly patients with ovarian, primary peritoneal cavity, or fallopian tube cancer | Up to 5 years
Percent of patients reporting adverse events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events | Up to 6 weeks after course 4
  The probability of an adverse event will be estimated as the percent of patients reporting an adverse event out of all patients beginning treatment.

OTHER OUTCOMES:
Pharmacokinetic parameters including paclitaxel AUC, carboplatin AUC, paclitaxel total body clearance, and time that plasma paclitaxel concentration remains above threshold 0.05 uM/L | Pre-dose, 1, 6, and 24 hours
  The observed pharmacokinetics of paclitaxel and carboplatin will be compared with published pharmacokinetic measures of paclitaxel and carboplatin in a descriptive fashion. No formal statistical testing will be performed for the comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian E von Gruenigen, Principal Investigator — Gynecologic Oncology Group
Locations (357):
- United States (357):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mercy Hospital, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Beth Israel Deaconess Hospital-Plymouth, Plymouth, Massachusetts
  - UMass Memorial Medical Center - Memorial Division, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Park Nicollet Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic-Tulsa South, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming